CLINICAL TRIAL: NCT06274827
Title: Electromyographic Analysis of Scapular Muscles During Closed Kinetic Chain Exercises: The Effect of Glenohumeral Joint Elevation Status on Muscle Activity
Brief Title: Electromyographic Analysis of Scapular Muscles During Closed Kinetic Chain Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Elif Turgut, Associate Professor Elif TURGUT, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GO 22- 881
Record Dates: First submitted 2024-02-01; First posted 2024-02-23 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Shoulder Pain; Shoulder Injuries; Activation, Patient
Keywords: Scapular muscle; Exercise; Electromyography; Kinetic chain
MeSH Terms: conditions — Shoulder Pain; Shoulder Injuries; Patient Participation; Motor Activity

STUDY DESIGN:
Intervention Model Description: All participants will complete each stage in a randomized order.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Superficial electromyography (Experimental): Electrode placement was performed on the participants' dominant side UT, MT, LT, and SA muscles. Following this, superficial electromyography measurements were performed during maximal voluntary isometric contraction tests and six different upper extremity closed kinetic chain exercises.
  Interventions: Diagnostic Test: Superficial Electromyography

INTERVENTIONS:
Diagnostic Test: Superficial Electromyography — For all MVICs, five seconds of each repetition were included in the analysis and the maximum value of three repetitions was taken. For all exercises, the middle 3 seconds of the 5 second data collection period were included in the analysis and the average muscle activation level of the three repetitions was recorded. The average signal amplitude of each exercise was divided by the MVIC of each muscle of interest to obtain the %MVIC value.
  Other Names: sEMG

SUMMARY:
In shoulder rehabilitation, the inclusion of kinetic chain exercises is advocated in order to provide the necessary energy transfer to produce optimal force with minimal energy consumption. Closed kinetic chain (CKC) exercises are defined as exercises in which the distal segment is stabilized by encountering significant resistance while the proximal segment moves. In contrast, open kinetic chain (OKC) exercises allow the distal segment to move freely without any resistance. Recently, the importance of closed kinetic chain (CKC) exercises has increased in enhancing shoulder joint neuromuscular control by improving dynamic shoulder stability and joint position sense.

The most current shoulder rehabilitation protocols include exercises for restoration of scapular muscle imbalances.There exist studies investigating the levels of scapular muscle activation during CKC exercises. Researchers have shown that most CKC exercises especially push-ups and plank variations with the shoulder in the 90° position, generally provide high SA activity and an optimal UT/SA ratio.In the literature, there is limited information on how the level of shoulder elevation affects scapular muscle activity and ratio during closed kinetic chain exercises in the prone position. To effectively prescribe CKC exercises commonly used in rehabilitation and athletic programs, a clear understanding of shoulder elevation changes muscle activity during these exercises is required.

Our hypothesis is that glenohumeral joint elevation status will alter scapular muscle activation and activation rates.

DETAILED DESCRIPTION:
Twenty-two healthy male individuals to recruited in the study. Conducting a power analysis through G∗Power, considering a moderate effect size (f = 0.25), an alpha level of 0.05, and a power of 0.8. The outcome of this analysis indicated a required minimum sample size of 21 individuals. This study was used a randomized, repeated measures cross-over design. Muscle activation levels during maximum voluntary isometric contraction (MVIC) of each muscle (Upper trapezius, Middle trapezius, Lower trapezius, Serratus anterior) will be recorded to normalize muscle activation levels during closed kinetic chain exercises. Muscle activation levels will be evaluated with a surface electromyography device (Noraxon, Myomotion, USA).

ELIGIBILITY:
Inclusion Criteria:

* Physically active male individuals (self-reported participating in 150 minutes per week of moderate-vigorous aerobic activity)
* Being between 18-30 years old
* Having full range of motion of shoulder without pain
* Having a body mass index less than 30 kg\m2.

Exclusion Criteria:

* Having pain in any kinetic chain of the body, had history of any musculoskeletal problems or orthopaedic surgery,
* Having symptoms in at least one of the screening tests (Hawkins-Kennedy, Neer, Resistant External Rotation, Jobe and Apprehension Test),
* Being diagnosed with a rheumatic, systemic or neurological disease.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy, physically active
Enrollment: 22 (Actual)
Dates: Start 2022-09-25 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Muscle activation recorded with surface electromyography (sEMG) during CKC | 2 hours for each participant
  In this study, muscle activations of the Upper Trapezius (UT), Middle Trapezius (MT), Lower Trapezius (LT), and Serratus Anterior (SA) muscles during six different closed kinetic chain (CKC) exercises will be investigated. The exercises include Low Plank Plus, High Plank Plus, Stir the Pot, Body Saw, Dolphin Press, and Pike Press. The average signal amplitude of each exercise will be divided by the Maximum Voluntary Isometric Contraction (MVIC) of each muscle of interest to obtain the %MVIC value. The average %MVICs will also be used for UT/MT, UT/LT, and UT/SA ratio calculations.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No